CLINICAL TRIAL: NCT02389166
Title: Randomized Clinical Trial Comparing High Flow Oxygen Delivery System (Optiflow) With Oxygen Therapy Under High-concentration Mask on Oxygenation of Patients Who Receive Sequential Non-Invasive Ventilation (NIV) Sessions
Brief Title: Optiflow in Sequential Non-Invasive Ventilation
Acronym: VNI-HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2013/28
Record Dates: First submitted 2015-03-03; First posted 2015-03-17 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optiflow group (Experimental)
  Interventions: Device: Optiflow
- Control group (Active Comparator)
  Interventions: Device: Conventional oxygen therapy

INTERVENTIONS:
Device: Optiflow — Patients receive high flow oxygen delivery system, Optiflow, conventional clinical management and sequential used of NIV for a period of 36 hours at least.
  High flow oxygen nasal therapy (Optiflow) : The flow will be set at 40l/min to 60l/min The inspired fraction of oxygen (FiO2) is the same as that defined at the end of VNI session and may be adjusted in order to obtain a SaO2 between 94% and 98%.
  Arms: Optiflow group
Device: Conventional oxygen therapy — Patients receive conventional oxygen therapy with high concentration mask, conventional clinical management, and sequential use of NIV Conventional oxygen therapy: The inspired fraction of oxygen (FiO2) is the same as that defined at the end of VNI session and may be adjusted in order to obtain a Arterial Oxygen Saturation (SaO2) between 94% and 98%.
  Arms: Control group

SUMMARY:
Background : Patient with hypoxemic respiratory failure treated with NIV receive between NIV session oxygen therapy. Gaz exchange disorder with a decrease of the ratio between Partial Pressure of Arterial Oxygen (PaO2) and Inspired Fraction of Oxygen (FIO2) are noticed when NIV is stopped at the end of the session du to alveolar derecruitment Optiflow is a high flow oxygen delivery system used a heated humidifier and heated breathing circuit. In observational studies, Optiflow increase oxygenation of patients with hypoxemic respiratory failure. Oxygenation is better than under high-concentration mask and work of breathing is reduced.

The aim of the study is to compare in acute hypoxemic respiratory failure, optiflow to oxygen therapy under high-concentration mask, on patients oxygenation between NIV sessions (measured as the difference between PaO2/FiO2 ratio at the beginning and at the end of the session), during the first two NIV sessions

Study design : Prospective, randomized, controlled, multicentric, open clinical trial with two groups:

* control group with conventional clinical management, oxygen therapy and sequential used of NIV
* Optiflow group with high flow oxygen delivery system, conventional clinical management and sequential used of NIV for a period of 36 hours at least.

Number of subjects: 100 (50 patients per group) patients admitted in intensive Care Unit for hypoxemic respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years old
* Patients affiliated to or benefiting of the French social welfare system
* Patients with ARDS on previously healthy lung. Acute respiratory insufficiency, defined as the PaO2/FIO2 ratio less than 200 mm Hg associated with the presence of lung infiltrates on chest radiograph
* Free and informed consent of patient
* Hospitalized in one of involved ICU

Exclusion Criteria:

* Existence of criteria for intubation.
* Refusal to participate in the study.
* Pregnancy
* Patient under guardianship or trusteeship
* Patients for whom a decision of non intubation has been decided.
* Patients who have received one or several NIV session for ARDS before hospital admission
* Home noninvasive ventilation
* Tracheostomy
* Hemodynamic instability
* Hypercapnia (PaCO2>45 mm Hg).
* left ventricular failure (cardiogenic pulmonary acute edema).
* Ineffective coughing.
* Recent gastric or oesophageal surgery
* Severe ventricular rhythm disorder
* High digestive haemorrhage
* Lack of collaboration
* Pernicious vomiting
* Upper airway obstruction
* Severe sepsis.
* Undrained pneumothorax.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2015-06-25 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
Average of oxygenation differences measured as the delta between PaO2/FiO2ratio at the end of the first ans second NIV session and at the end of the first and second oxygen therapy session. | 28 days
  Average of oxygenation differences measured as the delta between PaO2/FiO2 ratio at the end of the first NIV session and at the end of the first oxygen therapy session (according group of treatment) on the one hand and on the other hand the delta between PaO2/FiO2 ratio at the end of the second NIV session and at the end of the second oxygen thrapy session
  Five measurements of PaO2/FiO2 ratio are realized with arterial blood gases:
  * at the time of inclusion,
  * at the time of the end of first NIV session,
  * at the time of the end of first oxygen therapy session, or at the time of rescue NIV or at the time of réintubation
  * at the time of the end of second NIV session,
  * at the time of the end of second oxygen therapy session These five measurements are usually realised, and they are important to optimize patient management. The primary endpoint is based on these five measurements.

SECONDARY OUTCOMES:
comfort score dyspnea beetween the two NIV sessions | 28 days
  The comfort score and dyspnea will be assessed between the two NIV sessions
Incidence of serious adverse events between the two NIV sessions | 28 days
Respiratory rate between the two NIV sessions | 28 days
  Respiratory rate to assess work of breathing between the two NIV sessions
incidence of intubation during the NIV treatment of Acute respiratory distress syndrome (ARDS) | 28 days
ICU mortality | 28 days
28 days survival | 28 days
Hospital mortality | 28 days
ICU length of stay | 28 days
duration of mechanical ventilation | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Antoine BENARD, Docotor, Study Chair — University Hospital, Bordeaux
Locations (8):
- France (8):
  - Service de réanimation - CH de la côte basque, Bayonne, Aquitaine
  - Service de réanimation médicale - CHU de Bordeaux, Bordeaux, Aquitaine
  - Service de Réanimation Polyvalente - CH de Libourne, Libourne, Aquitaine
  - Service de Réanimation - CH de Perigueux, Périgueux, Aquitiane
  - Service de Réanimation Polyvalente - CHU de Toulouse, Toulouse, Midi-pyrenees
  - Service de Réanimation Polyvalente - CH d'Agen, Agen
  - Réanimation polyvalente - CH d'Albi, Albi
  - Réanimation Polyvalente - CH de Mont de Marsan, Mont-de-Marsan

IPD SHARING:
Plan to Share IPD: No